CLINICAL TRIAL: NCT03371264
Title: Optimizing Donor-recipient Matching to Improve Survival After Registration on the Waiting List for Liver Transplantation: the OPTIMATCH LT Study
Brief Title: Data Collection Study From Donors and Recipients to Optimize Donor-recipient Matching in Liver Transplantation
Acronym: OPTIMATCH-LT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Other Study IDs: P13639
Record Dates: First submitted 2017-11-17; First posted 2017-12-13 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; Allocation process; Extended-criteria donors; Survival

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort R1 and Cohort T1: Cohort R1 (patients on the waiting list between 2009 and 2013) and Cohort T1 (transplanted patients between 2009 and 2013)
- Cohort R2 and Cohort T2: Cohort R2 (patients on the waiting list in 2014) and Cohort T2 (transplanted patients in 2014)

SUMMARY:
A major limitation of liver transplantation is organ shortage. To avoid exposing patients to death on the waiting list, organs are used that would have been discarded few years ago. Graft allocation is regulated by the "agence de biomedecine" which establishes a national score. Each liver graft is proposed to the patient presenting the higher score. Acceptance or rejection of the graft only depends on the decision of each centre. We propose to submit a more efficient allocation model (enabling each proposed liver graft to be transplanted in the candidate whose transplantation will afford the greatest survival benefit after registration), by collecting and analysing variables from donors and candidates/recipients.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplant candidates : All adult LT candidates listed on the French wait list between 2009 and 2014 and followed prospectively by the mean yearly follow-up under the control of ABM.
* Donors : all adults donors registered over the same 2009-2014 period, including donors whose livers were procured and transplanted, whose liver were procured and discarded, and donors in whom liver was not harvested.

Exclusion Criteria:

* Pediatric recipients
* Pediatric donors

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population of proposed donors and the population of patients registered on the national waiting list from 2009 to 2014 (Agence de Biomédecine)
Sampling Method: Non-Probability Sample
Enrollment: 9000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Survival analysis | 5 years
  In view of the complexity of our project, different parallel approaches will be performed in order to establish predictive models
Multi-state models | 5 years
  In view of the complexity of our project, different parallel approaches will be performed in order to establish predictive models
Decision tree analysis | 5 years
  In view of the complexity of our project, different parallel approaches will be performed in order to establish predictive models

SECONDARY OUTCOMES:
Number of each criterion of ECD (Donor population) | 5 years
Percentage of each criterion of ECD (Donor population) | 5 years
Donor scores (DRI, ELTR) (Donor population) | 5 years
mean score (Donor population) | 5 years
number of ECD criteria (Donor population) | 5 years
frequency of ECD criteria (Donor population) | 5 years
mean age of donors (Donor population) | 5 years
graft failure (Donor population) | 5 years
grafts with correct primary function (Donor population) | 5 years
epidemiological characteristics (Candidate population) | 5 years
indication for transplantation (Candidate population) | 5 years
severity of disease (Candidate population) | 5 years
comorbidities (Candidate population) | 5 years
time on waiting list (Candidate population) | 5 years
Proportion of early deaths after transplantation (Candidate population) | 5 years
drop-outs for worsening (Candidate population) | 5 years
  Description of events occurring on waiting list
deaths on the waiting list (Candidate population) | 5 years
median time of occurrence (Candidate population) | 5 years
  Description of events occurring on waiting list
number of drop-outs for improvement (Candidate population) | 5 years
percentages of drop-outs for improvement (Candidate population) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Feray, MD/PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No